CLINICAL TRIAL: NCT06049641
Title: Hypertension in High School Students: Genetic and Environmental Factors
Brief Title: Hypertension in High School Students
Acronym: HYGEF
Status: Completed | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Chiara Lanzani, professor of Nephrology, Ospedale San Raffaele
Other Study IDs: HYGEF STUDY
Record Dates: First submitted 2023-09-05; First posted 2023-09-22 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Hypertension in Adolescence; Adolescent Overweight
Keywords: hypertension; adolescence; obesity; genetic
MeSH Terms: conditions — Pediatric Obesity; Hypertension; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Saliva
  * concentrated DNA in biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 13 to 15 Year-Old: * Normotensive (Normal BP): SBP and/or DBP values below the 90th percentile for teens of the same age and sex.
  * Prehypertensive (High-normal BP): SBP and/or DBP values at or above the 90th percentile and/or below the 95th percentile for for teens of the same age and sex.
  * Hypertensive: SBP and/or DBP values at or above the 95th percentile for teens of the same age and sex.
- 16 to 19 Year-Old: * Normotensive (Normal BP): SBP <130 mmHg and/or DBP <85 mm Hg.
  * Prehypertensive (High-normal BP): SBP 130 to 139 mmHg and/or DBP 85 to 89 mm Hg.
  * Hypertensive: SBP ≥140 mm Hg and/or DBP ≥90 mmHg.

SUMMARY:
Hypertension and obesity in the young population are major risk factors for renal and cardiovascular events, which could arise in adulthood. A candidate-gene approach will be applied in a cohort observational study, in which investigators will collect data from high school adolescent students. Participants underwent anthropometric and blood pressure measurements, as well as saliva and urine sample collection for genomic DNA extraction and renal function evaluation, respectively. Candidate genes previously implicated in salt-sensitive hypertension in adults will be tested to verify impact on blood pressure (BP) also among adolescents. Since inflammatory mechanisms may be involved in pathophysiology of hypertension and in endothelial dysfunction and atherosclerosis through reactive oxygen species, the baseline urinary excretion of inflammatory and oxidative stress markers in a subgroup of adolescents stratified according to ADD1 (alpha adducin) rs4961 genotypes will be assessed.

DETAILED DESCRIPTION:
Pediatric hypertension is associated with cardiovascular organ damage, which in turn may lead to cardiovascular disease (CVD) and acute events in adulthood.1 Over the past few decades, the prevalence of hypertension has progressively increased in children and adolescents, generating a significant public health issue and considerable amount of research. BP values among adolescents tend to be less heterogeneous than in adults, and the impact of genetic factors, even if small, may be the expression of pathogenic mechanisms that have been present since birth.

With this study, named HYGEF (Hypertension in high school students: Genetic and Environmental Factors), authors wanted to: 1. determine the prevalence of obesity and hypertension (HT) in a cohort of adolescents, 2. perform genetic analyses to determine a link between specific polymorphisms and/or mutations of genes involved in the development of HT in adults like the Adducin genes and Endogenous Ouabain (EO) and HT and 3. explore whether urine Na+/K+ excretion and urinary markers of inflammation and oxidative stress are linked to HT and cardiovascular risk in participants with the selected genotypes.

Adolescents will be enrolled for the study in high schools in the north (Milan), center (Livorno) and south (Grottaglie) of Italy, to obtain a sample that could be representative of the italian adolescents. During the visit at the high school investigators obtain questionnaires to have some information about eating habits, lifestyle and family history, two (or three in they were very discordant) blood pressure measurements, weight and height of the students, a sample of urine and a sample of saliva to extract DNA.

Genotyping: On the basis of our previous genetic studies carried out in adult patients with hypertension and cardiovascular and renal related diseases, 15 SNPs located in 13 candidate genes have been selected: rs1045642 in ABCB1, rs4343 in ACE (angiotensin converting enzyme), rs4961 in ADD1 (alpha-adducin), rs4984 in ADD2 (beta-adducin), rs3731566 in ADD3 (gamma-adducin), rs11638442 in CYP11A1 (cytochrome P450 family 11 subfamily A member 1), rs1799998 in CYP11B2 (aldosterone synthase), rs2236780, rs6203 and rs10923835 in HSD3B1 genetic region, rs9536314 in KL, rs2254524 in LSS, rs4149601 in neural precursor cell expressed, developmentally down-regulated 4-like, NEDD4L (E3 ubiquitin-protein ligase), PRKG1 (protein kinase, rs1904694 in cGMP-dependent, type I), rs4238595 in UMOD (uromodulin).

Analysis of Urines: Na+, K+, albumin, and creatinine were measured on a first fasting morning urine sample. The Kawasaki formula was used to estimate 24-hour urinary sodium (24h UNa) excretion expressed as mEq/24 h. In a subgroup a urine spot sample for each student will be immediately frozen for protein analysis. Investigators plan to measure simultaneously IL1β, IL6, IL10, IL12p70, TNF-α, MCP1 (monocyte chemoattractant protein), PTX3 (pentraxin-3) by ELISA test using LXSAHM Human Magnetic Luminex Screening Assay. Soluble α- Klotho, 8-Oxo-2'-deoxyguanosine will be measured by Elisa kit assay. Nitric oxide (NO) was measured by the colorimetric Nitric Oxide Assay kit. Advanced Oxidation Protein Products will be measured using the colorimetric OxiSelect Advanced Oxidation Protein Products Assay Kit.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 and 19 years old
* Caucasian

Exclusion Criteria:

* Age more than 19 years old
* Not Caucasian

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The final sample included 2638 white adolescents, 56% were females, 30% were from Milano (North Italy), 44% from Livorno (central Italy), and 26% from Grottaglie (South Italy).
Sampling Method: Non-Probability Sample
Enrollment: 2638 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
The aim of the study was to establish a link of specific polymorphisms of Adducins and EO-related genes with selected phenotypes (hypertension, Na+ and K+ intake). | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Background] de Simone G, Devereux RB, Daniels SR, Koren MJ, Meyer RA, Laragh JH. Effect of growth on variability of left ventricular mass: assessment of allometric signals in adults and children and their capacity to predict cardiovascular risk. J Am Coll Cardiol. 1995 Apr;25(5):1056-62. doi: 10.1016/0735-1097(94)00540-7. PMID 7897116
- [Background] Lurbe E, Agabiti-Rosei E, Cruickshank JK, Dominiczak A, Erdine S, Hirth A, Invitti C, Litwin M, Mancia G, Pall D, Rascher W, Redon J, Schaefer F, Seeman T, Sinha M, Stabouli S, Webb NJ, Wuhl E, Zanchetti A. 2016 European Society of Hypertension guidelines for the management of high blood pressure in children and adolescents. J Hypertens. 2016 Oct;34(10):1887-920. doi: 10.1097/HJH.0000000000001039. PMID 27467768
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Intersalt: an international study of electrolyte excretion and blood pressure. Results for 24 hour urinary sodium and potassium excretion. Intersalt Cooperative Research Group. BMJ. 1988 Jul 30;297(6644):319-28. doi: 10.1136/bmj.297.6644.319. PMID 3416162
- [Background] Citterio L, Lanzani C, Manunta P, Bianchi G. Genetics of primary hypertension: the clinical impact of adducin polymorphisms. Biochim Biophys Acta. 2010 Dec;1802(12):1285-98. doi: 10.1016/j.bbadis.2010.03.014. Epub 2010 Apr 8. PMID 20382219
- [Background] Efendiev R, Krmar RT, Ogimoto G, Zwiller J, Tripodi G, Katz AI, Bianchi G, Pedemonte CH, Bertorello AM. Hypertension-linked mutation in the adducin alpha-subunit leads to higher AP2-mu2 phosphorylation and impaired Na+,K+-ATPase trafficking in response to GPCR signals and intracellular sodium. Circ Res. 2004 Nov 26;95(11):1100-8. doi: 10.1161/01.RES.0000149570.20845.89. Epub 2004 Nov 4. PMID 15528469
- [Background] Manunta P, Maillard M, Tantardini C, Simonini M, Lanzani C, Citterio L, Stella P, Casamassima N, Burnier M, Hamlyn JM, Bianchi G. Relationships among endogenous ouabain, alpha-adducin polymorphisms and renal sodium handling in primary hypertension. J Hypertens. 2008 May;26(5):914-20. doi: 10.1097/HJH.0b013e3282f5315f. PMID 18398333
- [Background] Ferrari P. Rostafuroxin: an ouabain-inhibitor counteracting specific forms of hypertension. Biochim Biophys Acta. 2010 Dec;1802(12):1254-8. doi: 10.1016/j.bbadis.2010.01.009. Epub 2010 Jan 18. PMID 20083196
- [Background] Blaustein MP, Chen L, Hamlyn JM, Leenen FH, Lingrel JB, Wier WG, Zhang J. Pivotal role of alpha2 Na+ pumps and their high affinity ouabain binding site in cardiovascular health and disease. J Physiol. 2016 Nov 1;594(21):6079-6103. doi: 10.1113/JP272419. Epub 2016 Jul 31. PMID 27350568
- [Background] Manunta P, Iacoviello M, Forleo C, Messaggio E, Hamlyn JM, Lucarelli K, Guida P, Romito R, De Tommasi E, Bianchi G, Rizzon P, Pitzalis MV. High circulating levels of endogenous ouabain in the offspring of hypertensive and normotensive individuals. J Hypertens. 2005 Sep;23(9):1677-81. doi: 10.1097/01.hjh.0000177049.38417.67. PMID 16093912
- [Background] Nzietchueng R, El Shamieh S, Benachour H, Labat C, Herbeth B, Ndiaye NC, Masson C, Visvikis-Siest S, Benetos A. Klotho KL-VS genotype is involved in blood pressure regulation. Clin Chim Acta. 2011 Sep 18;412(19-20):1773-7. doi: 10.1016/j.cca.2011.05.032. Epub 2011 Jun 1. PMID 21663735
- [Background] Zhou X, Chen K, Lei H, Sun Z. Klotho gene deficiency causes salt-sensitive hypertension via monocyte chemotactic protein-1/CC chemokine receptor 2-mediated inflammation. J Am Soc Nephrol. 2015 Jan;26(1):121-32. doi: 10.1681/ASN.2013101033. Epub 2014 Jun 5. PMID 24904083
- [Background] Manunta P, Lavery G, Lanzani C, Braund PS, Simonini M, Bodycote C, Zagato L, Delli Carpini S, Tantardini C, Brioni E, Bianchi G, Samani NJ. Physiological interaction between alpha-adducin and WNK1-NEDD4L pathways on sodium-related blood pressure regulation. Hypertension. 2008 Aug;52(2):366-72. doi: 10.1161/HYPERTENSIONAHA.108.113977. Epub 2008 Jun 30. PMID 18591455
- [Background] Citterio L, Simonini M, Zagato L, Salvi E, Delli Carpini S, Lanzani C, Messaggio E, Casamassima N, Frau F, D'Avila F, Cusi D, Barlassina C, Manunta P. Genes involved in vasoconstriction and vasodilation system affect salt-sensitive hypertension. PLoS One. 2011 May 9;6(5):e19620. doi: 10.1371/journal.pone.0019620. PMID 21573014
- [Background] Trudu M, Janas S, Lanzani C, Debaix H, Schaeffer C, Ikehata M, Citterio L, Demaretz S, Trevisani F, Ristagno G, Glaudemans B, Laghmani K, Dell'Antonio G; SKIPOGH team; Loffing J, Rastaldi MP, Manunta P, Devuyst O, Rampoldi L. Common noncoding UMOD gene variants induce salt-sensitive hypertension and kidney damage by increasing uromodulin expression. Nat Med. 2013 Dec;19(12):1655-60. doi: 10.1038/nm.3384. Epub 2013 Nov 3. PMID 24185693
- [Background] Kuznetsova T, Staessen JA, Thijs L, Kunath C, Olszanecka A, Ryabikov A, Tikhonoff V, Stolarz K, Bianchi G, Casiglia E, Fagard R, Brand-Herrmann SM, Kawecka-Jaszcz K, Malyutina S, Nikitin Y, Brand E; European Project On Genes in Hypertension (EPOGH) Investigators. Left ventricular mass in relation to genetic variation in angiotensin II receptors, renin system genes, and sodium excretion. Circulation. 2004 Oct 26;110(17):2644-50. doi: 10.1161/01.CIR.0000145541.63406.BA. Epub 2004 Oct 18. PMID 15492316
- [Background] Staessen JA, Wang JG, Brand E, Barlassina C, Birkenhager WH, Herrmann SM, Fagard R, Tizzoni L, Bianchi G. Effects of three candidate genes on prevalence and incidence of hypertension in a Caucasian population. J Hypertens. 2001 Aug;19(8):1349-58. doi: 10.1097/00004872-200108000-00002. PMID 11518842
- [Background] Tripodi G, Citterio L, Kouznetsova T, Lanzani C, Florio M, Modica R, Messaggio E, Hamlyn JM, Zagato L, Bianchi G, Staessen JA, Manunta P. Steroid biosynthesis and renal excretion in human essential hypertension: association with blood pressure and endogenous ouabain. Am J Hypertens. 2009 Apr;22(4):357-63. doi: 10.1038/ajh.2009.3. Epub 2009 Feb 5. PMID 19197249
- [Background] Munshi A, Sharma V, Kaul S, Rajeshwar K, Babu MS, Shafi G, Anila AN, Balakrishna N, Alladi S, Jyothy A. Association of the -344C/T aldosterone synthase (CYP11B2) gene variant with hypertension and stroke. J Neurol Sci. 2010 Sep 15;296(1-2):34-8. doi: 10.1016/j.jns.2010.06.013. Epub 2010 Jul 3. PMID 20598712
- [Background] Tanase DM, Gosav EM, Radu S, Ouatu A, Rezus C, Ciocoiu M, Costea CF, Floria M. Arterial Hypertension and Interleukins: Potential Therapeutic Target or Future Diagnostic Marker? Int J Hypertens. 2019 May 2;2019:3159283. doi: 10.1155/2019/3159283. eCollection 2019. PMID 31186952
- [Background] Li Y, Thijs L, Kuznetsova T, Zagato L, Struijker-Boudier H, Bianchi G, Staessen JA. Cardiovascular risk in relation to alpha-adducin Gly460Trp polymorphism and systolic pressure: a prospective population study. Hypertension. 2005 Sep;46(3):527-32. doi: 10.1161/01.HYP.0000174988.81829.72. Epub 2005 Jul 25. PMID 16043664
- [Background] Manunta P, Ferrandi M, Cusi D, Ferrari P, Staessen J, Bianchi G. Personalized Therapy of Hypertension: the Past and the Future. Curr Hypertens Rep. 2016 Mar;18(3):24. doi: 10.1007/s11906-016-0632-y. PMID 26915067
- [Background] Liu M, Li Y, Citterio L, Huang QF, Zeng WF, Sheng CS, Wei FF, Dong Q, Li GL, Kang YY, Zhang L, Xu TY, Li JJ, Song J, Manunta P, Wang JG. A functional common polymorphism of the ABCB1 gene is associated with chronic kidney disease and hypertension in Chinese. Am J Hypertens. 2013 Dec;26(12):1428-36. doi: 10.1093/ajh/hpt126. Epub 2013 Aug 7. PMID 23926124
- [Background] Seidlerova J, Staessen JA, Bochud M, Nawrot T, Casamassima N, Citterio L, Kuznetsova T, Jin Y, Manunta P, Richart T, Struijker-Boudier HA, Fagard R, Filipovsky J, Bianchi G. Arterial properties in relation to genetic variations in the adducin subunits in a white population. Am J Hypertens. 2009 Jan;22(1):21-6. doi: 10.1038/ajh.2008.261. Epub 2008 Sep 11. PMID 18787518
- [Background] Iatrino R, Lanzani C, Bignami E, Casamassima N, Citterio L, Meroni R, Zagato L, Zangrillo A, Alfieri O, Fontana S, Macrina L, Delli Carpini S, Messaggio E, Brioni E, Dell'Antonio G, Manunta P, Hamlyn JM, Simonini M. Lanosterol Synthase Genetic Variants, Endogenous Ouabain, and Both Acute and Chronic Kidney Injury. Am J Kidney Dis. 2019 Apr;73(4):504-512. doi: 10.1053/j.ajkd.2018.10.012. Epub 2019 Jan 16. PMID 30660405
- [Background] Citterio L, Ferrandi M, Delli Carpini S, Simonini M, Kuznetsova T, Molinari I, Dell' Antonio G, Lanzani C, Merlino L, Brioni E, Staessen JA, Bianchi G, Manunta P. cGMP-dependent protein kinase 1 polymorphisms underlie renal sodium handling impairment. Hypertension. 2013 Dec;62(6):1027-33. doi: 10.1161/HYPERTENSIONAHA.113.01628. Epub 2013 Sep 23. PMID 24060892
- [Background] Kawasaki T, Itoh K, Uezono K, Sasaki H. A simple method for estimating 24 h urinary sodium and potassium excretion from second morning voiding urine specimen in adults. Clin Exp Pharmacol Physiol. 1993 Jan;20(1):7-14. doi: 10.1111/j.1440-1681.1993.tb01496.x. PMID 8432042
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901
- [Background] Cappuccio FP, Ji C, Donfrancesco C, Palmieri L, Ippolito R, Vanuzzo D, Giampaoli S, Strazzullo P. Geographic and socioeconomic variation of sodium and potassium intake in Italy: results from the MINISAL-GIRCSI programme. BMJ Open. 2015 Sep 10;5(9):e007467. doi: 10.1136/bmjopen-2014-007467. PMID 26359282
- [Background] Welsh CE, Welsh P, Jhund P, Delles C, Celis-Morales C, Lewsey JD, Gray S, Lyall D, Iliodromiti S, Gill JMR, Sattar N, Mark PB. Urinary Sodium Excretion, Blood Pressure, and Risk of Future Cardiovascular Disease and Mortality in Subjects Without Prior Cardiovascular Disease. Hypertension. 2019 Jun;73(6):1202-1209. doi: 10.1161/HYPERTENSIONAHA.119.12726. PMID 31067194
- [Background] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Background] Andrukhova O, Slavic S, Smorodchenko A, Zeitz U, Shalhoub V, Lanske B, Pohl EE, Erben RG. FGF23 regulates renal sodium handling and blood pressure. EMBO Mol Med. 2014 Jun;6(6):744-59. doi: 10.1002/emmm.201303716. Epub 2014 Apr 6. PMID 24797667
- [Background] Cusi D, Barlassina C, Azzani T, Casari G, Citterio L, Devoto M, Glorioso N, Lanzani C, Manunta P, Righetti M, Rivera R, Stella P, Troffa C, Zagato L, Bianchi G. Polymorphisms of alpha-adducin and salt sensitivity in patients with essential hypertension. Lancet. 1997 May 10;349(9062):1353-7. doi: 10.1016/S0140-6736(97)01029-5. PMID 9149697
- [Background] Taylor WR. Hypertensive vascular disease and inflammation: mechanical and humoral mechanisms. Curr Hypertens Rep. 1999 Feb-Mar;1(1):96-101. doi: 10.1007/s11906-999-0079-5. PMID 10981048
- [Background] Libby P. Interleukin-1 Beta as a Target for Atherosclerosis Therapy: Biological Basis of CANTOS and Beyond. J Am Coll Cardiol. 2017 Oct 31;70(18):2278-2289. doi: 10.1016/j.jacc.2017.09.028. PMID 29073957
- [Background] Li QZ, Deng Q, Li JQ, Yi GH, Zhao SP. Valsartan reduces interleukin-1beta secretion by peripheral blood mononuclear cells in patients with essential hypertension. Clin Chim Acta. 2005 May;355(1-2):131-6. doi: 10.1016/j.cccn.2004.12.006. PMID 15820487
- [Background] Elijovich F, Weinberger MH, Anderson CA, Appel LJ, Bursztyn M, Cook NR, Dart RA, Newton-Cheh CH, Sacks FM, Laffer CL; American Heart Association Professional and Public Education Committee of the Council on Hypertension; Council on Functional Genomics and Translational Biology; and Stroke Council. Salt Sensitivity of Blood Pressure: A Scientific Statement From the American Heart Association. Hypertension. 2016 Sep;68(3):e7-e46. doi: 10.1161/HYP.0000000000000047. Epub 2016 Jul 21. No abstract available. PMID 27443572
- [Background] Lin RC, Morris BJ. Association analysis of polymorphisms at the interleukin-1 locus in essential hypertension. Am J Med Genet. 2002 Feb 1;107(4):311-6. doi: 10.1002/ajmg.10177. PMID 11840488
- [Background] Saraiva M, O'Garra A. The regulation of IL-10 production by immune cells. Nat Rev Immunol. 2010 Mar;10(3):170-81. doi: 10.1038/nri2711. Epub 2010 Feb 15. PMID 20154735
- [Background] Caligiuri G, Rudling M, Ollivier V, Jacob MP, Michel JB, Hansson GK, Nicoletti A. Interleukin-10 deficiency increases atherosclerosis, thrombosis, and low-density lipoproteins in apolipoprotein E knockout mice. Mol Med. 2003 Jan-Feb;9(1-2):10-7. PMID 12765335
- [Background] Lima VV, Zemse SM, Chiao CW, Bomfim GF, Tostes RC, Clinton Webb R, Giachini FR. Interleukin-10 limits increased blood pressure and vascular RhoA/Rho-kinase signaling in angiotensin II-infused mice. Life Sci. 2016 Jan 15;145:137-43. doi: 10.1016/j.lfs.2015.12.009. Epub 2015 Dec 9. PMID 26682936
- [Background] Chatterjee P, Chiasson VL, Seerangan G, Tobin RP, Kopriva SE, Newell-Rogers MK, Mitchell BM. Cotreatment with interleukin 4 and interleukin 10 modulates immune cells and prevents hypertension in pregnant mice. Am J Hypertens. 2015 Jan;28(1):135-42. doi: 10.1093/ajh/hpu100. Epub 2014 Jun 6. PMID 24906486
- [Background] Appel LJ, Brands MW, Daniels SR, Karanja N, Elmer PJ, Sacks FM; American Heart Association. Dietary approaches to prevent and treat hypertension: a scientific statement from the American Heart Association. Hypertension. 2006 Feb;47(2):296-308. doi: 10.1161/01.HYP.0000202568.01167.B6. PMID 16434724
- [Background] van den Hoogen PC, Feskens EJ, Nagelkerke NJ, Menotti A, Nissinen A, Kromhout D. The relation between blood pressure and mortality due to coronary heart disease among men in different parts of the world. Seven Countries Study Research Group. N Engl J Med. 2000 Jan 6;342(1):1-8. doi: 10.1056/NEJM200001063420101. PMID 10620642
- [Background] Jin Y, Kuznetsova T, Citterio L, Thijs L, Messaggio E, Casamassima N, Manunta P, Fagard R, Bianchi G, Staessen JA. Left ventricular structure and function in relation to steroid biosynthesis genes in a white population. Am J Hypertens. 2012 Sep;25(9):986-93. doi: 10.1038/ajh.2012.69. Epub 2012 Jun 7. PMID 22673022
- [Background] Tentori S, Messaggio E, Brioni E, Casamassima N, Simonini M, Zagato L, Hamlyn JM, Manunta P, Lanzani C. Endogenous ouabain and aldosterone are coelevated in the circulation of patients with essential hypertension. J Hypertens. 2016 Oct;34(10):2074-80. doi: 10.1097/HJH.0000000000001042. PMID 27457665
- [Background] Cooper RS, Zhu X. Racial differences and the genetics of hypertension. Curr Hypertens Rep. 2001 Feb;3(1):19-24. doi: 10.1007/s11906-001-0073-z. PMID 11177703
- [Background] Polonia J, Lobo MF, Martins L, Pinto F, Nazare J. Estimation of populational 24-h urinary sodium and potassium excretion from spot urine samples: evaluation of four formulas in a large national representative population. J Hypertens. 2017 Mar;35(3):477-486. doi: 10.1097/HJH.0000000000001180. PMID 27898506